CLINICAL TRIAL: NCT02021929
Title: Sorafenib in Patients With Hepatopulmonary Syndrome: A Double-Blind Randomized Clinical Trial
Brief Title: Sorafenib for Hepatopulmonary Syndrome
Acronym: SHPS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 819185; UM1HL116886 (NIH)
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Hepatopulmonary Syndrome
Keywords: Randomized Controlled Trial; Clinical Trial; sorafenib; Hepatopulmonary Syndrome
MeSH Terms: conditions — Hepatopulmonary Syndrome | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Experimental): 400 mg (2 capsules) taken by mouth once a day
  Interventions: Drug: Sorafenib
- Placebo (Placebo Comparator): 2 capsules taken by mouth once a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib — Sorafenib is a kinase inhibitor indicated for the treatment of:
  * Unresectable hepatocellular carcinoma
  * Advanced renal cell carcinoma
  * Locally recurrent or metastatic, progressive, differentiated thyroid carcinoma refractory to radioactive iodine treatment
  Other Names: Nexavar
  Arms: Sorafenib
Drug: Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this clinical trial is to determine the safety and effects of the study drug, sorafenib, in adults diagnosed with hepatopulmonary syndrome (HPS). The study will evaluate how well the drug is tolerated and its effect on the level of oxygen in the blood and the function of the lung vessels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HPS:

  1. AaPO2 ≥ 15 mm Hg (≥ 20 mm Hg for age > 64 yrs)
  2. Intrapulmonary shunting
  3. Absence of significant restriction (TLC < 70%) or obstruction (FEV1 < 80% & FEV1/FVC < 70%)
  4. Presence of cirrhosis/hepatic fibrosis and/or portal hypertension
* Child-Pugh class A or B liver disease
* Platelet count ≥ 30 ×10e9 per liter
* Hemoglobin ≥ 8.5 g per deciliter
* International normalized ratio ≤ 2.3
* Albumin ≥ 2.8 g per deciliter
* Total bilirubin ≤ 5 mg per deciliter
* Alanine aminotransferase and aspartate aminotransferase ≤ 5 times the upper limit of the normal range
* Serum creatinine ≤ 1.5 times the upper limit of the normal range and not receiving dialysis
* Negative pregnancy test (for women of childbearing potential) at both screening and baseline visits. Post-menopausal women (defined as no menses for one year) and surgically sterilized women are not required to undergo a pregnancy test.
* Subjects (men and women) of childbearing potential must agree to use medically acceptable contraception beginning at the signing of the Informed Consent Form until at least 14 days after the last dose of study drug.
* Age ≥ 21 years
* Ability to provide informed consent

Exclusion Criteria:

* Recent chronic heavy alcohol consumption
* Enrollment in a clinical trial or concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 28 days of screening visit
* Current hepatic encephalopathy
* Active infection
* Diagnosis of portopulmonary hypertension
* WHO Class IV functional status
* Congenital long-QT syndrome
* Subjects who have used strong CYP3A4 inducers (e.g., phenytoin, carbamazepine, phenobarbital, St. John's Wort [Hypericum perforatum], dexamethasone at a dose of greater than 16 mg daily, or rifampin [rifampicin], and/or rifabutin) within 28 days before randomization
* Subjects who are currently taking Coumadin®(warfarin)
* Active or clinically significant cardiac disease, including:

  1. Active coronary artery disease
  2. Unstable angina (anginal symptoms at rest), new-onset angina within 12 weeks before randomization, or myocardial infarction within 24 weeks before randomization
* Liver or other solid organ transplant recipients
* Expectation of liver transplant within four months of randomization
* Hepatocellular carcinoma that does not meet all of the following criteria:

  1. Single lesion ≤ 3 cm documented by LIRADS criteria
  2. Complete response to ablative therapy (TACE, RFA, alcohol ablation) using the modified RECIST criteria one month after therapy with no more than two treatments
  3. No other lesions develop after initiation of HCC therapy
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg on repeated measurement) despite optimal medical management.
* Any hemorrhage/bleeding event of NCI-Common Toxicity Criteria for Adverse Effects v4.0 Grade 3 or higher within 4 weeks before randomization
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* Women who are pregnant or breast-feeding
* Major surgery 28 days prior to randomization
* Subjects with any previously untreated or concurrent cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before randomization are allowed. All cancer treatments (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form).
* Inability to comply with the protocol and/or not willing or not available for follow-up assessments

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Kawut, MD, MS, Principal Investigator — University of Pennsylvania
Locations (7):
- United States (7):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Columbia University-NewYork-Presbyterian Hospital, New York, New York
  - University of Pennsylvania - Perelman Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center at Houston Medical School, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib: 400 mg (2 capsules) taken by mouth once a day
  Sorafenib: Sorafenib is a kinase inhibitor indicated for the treatment of:
  * Unresectable hepatocellular carcinoma
  * Advanced renal cell carcinoma
  * Locally recurrent or metastatic, progressive, differentiated thyroid carcinoma refractory to radioactive iodine treatment
- Placebo: 2 capsules taken by mouth once a day
  Placebo
Period: Overall Study
Arm/Group | Sorafenib | Placebo
Started | 16 | 12
Completed | 14 | 11
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib | Placebo | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [53 to 64] | 59 [54 to 63] | 60 [53 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 15 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 10 | 26
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 28
World Health Organization functional class [Count of Participants; unit: Participants] — Classification based on evaluation of the participant.
  Class I: Patients without limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain or near-syncope.
  Class II: Patients with slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain or near-syncope.
  Class III: Patients with marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes undue dyspnea or fatigue, chest pain or near-syncope.
  Participants
    Class I | 3 | 4 | 7
    Class II | 6 | 2 | 8
    Class III | 7 | 6 | 13
Childs-Pugh Class [Count of Participants; unit: Participants] — Child-Pugh Class consists of five clinical features and is used to assess the prognosis of chronic liver disease and cirrhosis. There are three distinct classes of increasing severity (A, B and C). Class is determined based on a score that accounts for five factors: total bilirubin level, serum albumin, INR, degree of ascites, and degree of hepatic encephalopathy.
  Participants
    A | 7 | 3 | 10
    B | 9 | 9 | 18
Model for End-stage Liver Disease [Median (Inter-Quartile Range); unit: units on a scale] — A numerical scale, ranging from 6 (less ill) to 40 (gravely ill), used for liver transplant candidates. It gives each person a number based on how urgently he or she needs a liver transplant within the next three months. The number is calculated by a formula using three routine lab test results:
  * bilirubin, which measures how effectively the liver excretes bile;
  * INR (prothrombin time), which measures the liver's ability to make blood clotting factors; and
  * creatinine, which measures kidney function. (Impaired kidney function is often associated with severe liver disease.)
  units on a scale | 13 [11 to 14] | 13 [10 to 15] | 13 [10 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Change in Alveolar-arterial Oxygen Gradient Between Sorafenib and Placebo Groups
Description: Alveolar-arterial oxygen gradient is a calculated measure of oxygenation. It is the difference between the amount of the oxygen in the alveoli and the amount of oxygen in arterial blood.
  Calculation is based on values from an Arterial Blood Gas test. Difference in change in alveolar-arterial oxygen gradient between sorafenib and placebo from baseline to 12 weeks.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 14 | 11
mm Hg | 4.5 [-3.8 to 7.0] | -2.4 [-4.8 to 8.2]

2. Secondary Outcome: Number of Participants With Improvement in Intrapulmonary Shunting From Baseline to 12 Weeks.
Description: Intrapulmonary shunting is measured based on results from a saline-bubble echo test.
  Number of participants with measured improvement in intrapulmonary shunting from baseline to 12 weeks in the sorafenib and placebo groups
Time Frame: Baseline to 12 weeks
Population: Since all of the participants did not complete the 12 week study visit, data from fewer participants were available to be analyzed in each arm for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 12 | 9
Participants | 3 | 6

3. Secondary Outcome: Change From Baseline in Percentage of Progenitor Cells (Peripheral Blood Mononuclear Cells or PBMCs)
Description: Progenitor Cells (Peripheral Blood Mononuclear Cells or PBMCs) are obtained and measured from blood samples collected from each participant.
  Difference in change from baseline to 12 weeks in the Percentage of Progenitor Cells between sorafenib and placebo groups.
Time Frame: Baseline to 12 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of PBMCs
Arm/Group | Sorafenib | Placebo
Number analyzed (Participants) | 12 | 10
percentage of PBMCs | 0.01 [-0.02 to 0.04] | 0.04 [0.00 to 0.07]

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Sorafenib | Placebo
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 7/16 | 5/12
Other Adverse Events (participants affected / at risk) | 16/16 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=16) | Placebo (N=12)
Encephalopathy (Hepatobiliary disorders) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Diagnostic procedure (General disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Liver transplant (Surgical and medical procedures) | 1 | 2
Platelet count low (Blood and lymphatic system disorders) | 0 | 1
Skin infection (Fournier's gangrene) (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=16) | Placebo (N=12)
Diarrhea (Gastrointestinal disorders) | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Weight loss (General disorders) | 5 | 2
Fatigue (General disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 3 | 3
Pruritus (General disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypertension (Cardiac disorders) | 3 | 2
Rash (maculo-papular) (Skin and subcutaneous tissue disorders) | 4 | 1
Headache (General disorders) | 4 | 0
Myalgia (General disorders) | 2 | 2
Alopecia (General disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Edema (Cardiac disorders) | 2 | 1
Mucositis (oral) (General disorders) | 3 | 0
Nasal congestion (General disorders) | 1 | 2
Pain in extremity (General disorders) | 2 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Recruitment difficult due to challenges in screening for HPS, lack of patient awareness of HPS, and hesitation from potential subjects due to sorafenib side effects. Sample size reduced and sponsor terminated trial before reaching target sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT02021929/Prot_SAP_000.pdf